CLINICAL TRIAL: NCT04679506
Title: Clinical Observation on the Efficacy and Safety of CLAE Regimen (Cladribine + Cytarabine + Etoposide) in the Treatment of Relapsed/Refractory T- Acute Lymphoblastic Leukemia/Lymphoblastic Lymphoma
Brief Title: the Efficacy and Safety of CLAE in R/R T-ALL/LBL
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CLAE
Record Dates: First submitted 2020-12-13; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Precursor T-Cell Lymphoblastic Leukemia-Lymphoma
Keywords: R/R T-ALL/LBL; CLAE
MeSH Terms: conditions — Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cladribine; Cytarabine; Etoposide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cladribine — CLAE regimen (cladribine + cytarabine + etoposide) for reinduction of R/R T-ALL/LBL
  Other Names: cytarabine; etoposide

SUMMARY:
To evaluate the efficacy and safety of CLAE regimen (cladribine + cytarabine + etoposide) in the treatment of relapsed/refractory T-ALL/LBL.

DETAILED DESCRIPTION:
This study is a prospective, open, multiple -centered, sing-arm trial. The major aim of this studies to evaluate the efficacy and safety of CLAE regimen (cladribine + cytarabine + etoposide) in the treatment of relapsed/refractory T-ALL/LBL. The study will include 50 subjects to receive CLAE regimen for reinduction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T-acute lymphoblastic leukemia/lymphoblastic lymphoma according to World Health Organization (WHO) criteria which has relapsed or is refractory to chemotherapy.
* Age ≥ 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* The expected survival period is more than 12 weeks.
* At least one measurable nidus
* Adequate organ function defined as:

  * Calculated creatinine clearance ≥ 50 ml/min using the cockcroft -Gault formula
  * AST, ALT, total bilirubin ≤ 2 x upper limit of normal (ULN) except for Gilbert's disease or when in the opinion of treating physician elevated levels are due to direct involvement of leukemia (e.g., hepatic infiltration or biliary obstruction due to leukemia), in which case ALT and AST may be elevated up to ≤ 5 x ULN.
* Able to understand and willing to sign an Institutional Review Board (IRB)-approved written informed consent document.

Exclusion Criteria:

* Previous treatment with nelarabine or clofarabine or fludarabine or cladribine was ineffective.
* Pregnant or nursing.
* Received any other investigational agent or systemic cytotoxic chemotherapy within the preceding 2 weeks.
* Active HIV or hepatitis B or C infection.
* Any medical condition which, in the opinion of the clinical investigator, would interfere with the evaluation of the patient. Subjects with a clinically significant or unstable medical or surgical condition or any other condition that cannot be well-controlled by the allowed medications permitted in the study protocol that would preclude safe and complete study participation, as determined by medical history, physical examinations, laboratory tests, and according to the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A singe-arm of patients with R/R T-ALL/LBL
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
ORR | From the date of first study drug administration until the end of Cycle 2 (each cycle is 28 days)
  Objective response rate，sum of complete response rate and partial response rate

SECONDARY OUTCOMES:
PFS | From the date of first study drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.
  progression-free survival
OS | From the date of first study drug administration until the date of death due to any cause, assessed up to 24 months.
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Hongmei Jing, MD, phD, Study Director — Peking University Third Hospital